CLINICAL TRIAL: NCT05908799
Title: Emulation of a Comparative Effectiveness Study of Pembrolizumab and Chemotherapy vs. Chemotherapy for the First-line Treatment of Metastatic Non-small Cell Lung Cancer
Brief Title: Emulation of the KEYNOTE-189 Trial Using Electronic Health Records
Status: Completed | Type: Observational
Sponsor: Aetion, Inc. (Other)
Responsible Party: Principal Investigator, David Merola, Principal Scientist, Aetion, Inc.
Other Study IDs: 1
Record Dates: First submitted 2023-06-07; First posted 2023-06-18 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Non-small Cell Lung Cancer; Metastatic Lung Cancer
Keywords: real-world evidence; real-world data; oncology; pharmacoepidemiology; comparative effectiveness research
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Pembrolizumab + Chemotherapy: Exposure Group
  Interventions: Drug: Pembrolizumab + Pemetrexed-Platinum
- Chemotherapy: Reference Group
  Interventions: Drug: Pemetrexed-Platinum

INTERVENTIONS:
Drug: Pembrolizumab + Pemetrexed-Platinum — Medication records in EHR database used to define exposure group
  Groups: Pembrolizumab + Chemotherapy
Drug: Pemetrexed-Platinum — Medication records in EHR database used to define comparator group
  Groups: Chemotherapy

SUMMARY:
Investigators are building an empirical evidence base supporting the utility of real-world data through the emulation of randomized controlled trials in the oncology setting. The purpose of this work is to demonstrate whether real-world evidence studies can provide reliable conclusions on treatment effectiveness to inform further applications of real-world data in pharmaceutical product label expansion, post-marketing safety, and other purposes that are complementary to RCTs.

DETAILED DESCRIPTION:
This is a non-randomized observational study that is being conducted as a part of the Coalition to Advance Real-World Evidence through Randomized Controlled Trial Emulation (CARE) Initiative, a multi-stakeholder collaboration led by Aetion. The study is intended to emulate the trial listed below/above. Although many features of the trial cannot be directly replicated in real-world data sources, key elements of the study design, including outcomes, exposures, and inclusion/exclusion criteria, were selected to proxy those features from the trial as closely as possible. Investigators assume that the trial provides the reference standard treatment effect estimate and that failure to replicate trial findings is indicative of the inadequacy of the real-world data source for replication for a range of possible reasons and does not provide information on the validity of the original trial finding.

ELIGIBILITY:
Inclusion Criteria:

* Has evidence in electronic health record indicating a 'lung' tumor site, non-squamous morphology (e.g., adenocarcinoma, large cell, etc), and a stage IV or metastatic disease in the form of diagnosis codes or derived variables from physician notes or linked data from a tumor registry. There is no evidence of other lung cancer types (i.e., mesothelioma, small cell, etc.).
* Does not have evidence of HGVS codes in health record indicating EGFR or ALK mutations.
* Has no evidence of use of guideline-recommended systemic cancer therapy* for NSCLC on or after first date associated with stage IV (or metastatic) disease and prior to index treatment.

Exclusion Criteria:

* Has evidence of squamous cell lung cancer morphology in the form of diagnosis codes or derived variables from physician notes or linked information from a tumor registry.
* Has evidence of systemic cancer therapy utilization on or after first date associated with stage IV (or metastatic) disease and prior to index treatment. Patient has no evidence of biologic therapy at any time prior to the first record indicating an exposure of interest.
* Has evidence in medical record or tumor registry of primary malignancies beyond the lung tissue, except basal cell carcinoma of the skin, superficial bladder cancer, squamous cell carcinoma of the skin, in situ cervical cancer, or other in situ cancers.
* Has evidence of central nervous system (CNS) metastases and/or carcinomatous meningitis in the 2 weeks prior to initiation.
* Has a record of use of one of the following agents in the 2 years prior to the index date: methotrexate, sulfasalazine, hydroxychloroquine, leflunomide, azathioprine, etanercept, adalimumab, infliximab, certolizumab, golimumab, anakinra, tocilizumab, sarilumumab, abatacept, rituximab, tofacitinib, barivitinib, upadacitinib, mycophenolate.
* Has at least two records 60 days apart indicating use of one of the following agents in the 3 months prior to the index date: prednisone, prednisolone, methylprednisolone, dexamethasone, hydrocortisone.
* Has evidence of use of one of the following agents prior to the index date: pembrolizumab, nivolumab, cemiplimab, atezolizumab, durvalumab.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Non-small cell lung cancer patients with evidence of metastatic disease and a subsequent record indicating a first-line treatment.
Sampling Method: Non-Probability Sample
Enrollment: 1854 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Overall Survival - Mortality Hazard Ratio | Through study completion (earliest of 640 days or censoring)
  Relative hazard of mortality due to any cause
Overall Survival - Mortality Risk | 1 year, year 1
  12-month survival probability

CONTACTS AND LOCATIONS:
Overall Officials: David Merola, PharmD, PhD, Principal Investigator — Aetion, Inc.
Locations (1):
- Aetion, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided
Data analysis code and de-identified patient-level data files may be made available, provided that it is determined that this will not violate the investigators' data usage agreements and patient privacy requirements.

REFERENCES:
- [Background] Merola D, Campbell U, Gautam N, Rubens A, Schneeweiss S, Wang SV, Carrigan G, Chia V, Ovbiosa OE, Pinheiro S, Bruno A, Jiao X, Stewart M, Hendricks-Sturrup R, Rodriguez-Watson C, Khosla S, Zhang Y, Rimawi M, Huang J, Taylor A, Becnel L, McRoy L, Eckert J, Taylor B. The Aetion Coalition to Advance Real-World Evidence through Randomized Controlled Trial Emulation Initiative: Oncology. Clin Pharmacol Ther. 2023 Jun;113(6):1217-1222. doi: 10.1002/cpt.2800. Epub 2022 Dec 7. PMID 36408668

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-09-08): https://cdn.clinicaltrials.gov/large-docs/99/NCT05908799/Prot_SAP_002.pdf